CLINICAL TRIAL: NCT00249457
Title: A Therapeutic Workplace for Drug Abusers
Brief Title: Employment-based Reinforcement to Motivate Drug Abstinence in the Treatment of Drug Addiction. - 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-13107-2
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Behavior, Addictive; Cocaine Abuse; Cocaine Dependence; Heroin Dependence; Opioid Dependence
Keywords: Behavior Therapy; Cocaine Abuse; Cocaine Dependence; Contingency Management; Heroin Dependence; Methadone; Opioid Dependence
MeSH Terms: conditions — Behavior, Addictive; Cocaine-Related Disorders; Heroin Dependence; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Workplace (Experimental): Contingency management. Invited to work in the Therapeutic Workplace. Completed monthly assessments.
  Interventions: Behavioral: Contingency management
- Usual Care Control Group (No Intervention): No intervention. Not invited to work int the Therapeutic Workplace. Completed monthly assessments.

INTERVENTIONS:
Behavioral: Contingency management — Invited to attend the Therapeutic Workplace 3 hr per day, Monday through Friday. Each day when a participant reported to the workplace, she was required to provide a urine sample. If the sample tested negative for opiates and cocaine, she was allowed to work that day. Participants who gained entrance to the workplace participated in basic skills education and job skills training throughout each 3-hr work shift.
  Arms: Therapeutic Workplace

SUMMARY:
The purpose of this study is to determine whether long-term exposure to the Therapeutic Workplace intervention could sustain drug abstinence over an extended period of time in heroin- and cocaine-dependent, unemployed, treatment-resistant young mothers.

DETAILED DESCRIPTION:
The current study is a continuation of the research into the development and evaluation of a novel treatment designed to address the chronic, persistent nature of drug addiction. This treatment, called the Therapeutic Workplace, integrates abstinence reinforcement contingencies of proven efficacy into a model supported work program. Participants were paid to work or to train in the Therapeutic Workplace but had to provide drug-free urine samples to gain daily access. Forty participants were randomly assigned to a Therapeutic Workplace or usual care control group. Therapeutic Workplace participants could work for about 5 years. This study reports the effects of the intervention over a follow-up period of 8 years after treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* When originally enrolled in the study, participants were at least 18 years old, unemployed, and methadone maintenance patients of the Center for Addiction and Pregnancy (CAP) who continued to use opiates or cocaine during CAP treatment.

Exclusion Criteria:

* Participants were excluded if they were at risk for suicide at the time of intake or if they had serious psychiatric illness (e.g., schizophrenia).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 1996-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Percentage of urine samples at the assessments that were negative for cocaine | every 30 days throughout fourth year
  (total number of monthly urine samples negative for cocaine/total number of possible urine samples) x 100
Percentage of urine samples at the assessments that were negative for opiates | every 30 days throughout fourth year
  (total number of monthly urine samples negative for opiates/total number of possible urine samples) x 100
Percentage of urine samples at the assessments that were negative for cocaine and opiates | every 30 days throughout fourth year
  (total number of monthly urine samples negative for cocaine and opiates/total number of possible urine samples) x 100

SECONDARY OUTCOMES:
HIV risk behaviors | every 30 days throughout fourth year
Percentage of participants employed each month | every 30 days throughout fourth year
Number of days employed each month | every 30 days throughout fourth year
Percentage of participants to self-report abstinence at all time points | every 30 days throughout fourth year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The data for this study have been published in a peer-reviewed journal.

REFERENCES:
- [Result] Aklin WM, Wong CJ, Hampton J, Svikis DS, Stitzer ML, Bigelow GE, Silverman K. A therapeutic workplace for the long-term treatment of drug addiction and unemployment: eight-year outcomes of a social business intervention. J Subst Abuse Treat. 2014 Nov-Dec;47(5):329-38. doi: 10.1016/j.jsat.2014.06.013. Epub 2014 Jul 12. PMID 25124257